CLINICAL TRIAL: NCT05681481
Title: An Open-label Extension Study of ARGX-113-2009 to Evaluate the Long Term Safety, Tolerability, and Efficacy of Efgartigimod PH20 SC in Adult Participants With Bullous Pemphigoid
Brief Title: A Phase 3 Study to Evaluate the Long-term Safety, Tolerability and Efficacy of Efgartigimod PH20 SC in Adult Participants With Bullous Pemphigoid
Acronym: BALLAD+
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARGX-113-2010; 2024-515832-59-00 (EU CTIS Number)
Record Dates: First submitted 2022-12-08; First posted 2023-01-12 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Bullous Pemphigoid
MeSH Terms: conditions — Pemphigoid, Bullous | interventions — Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- efgartigimod PH20 SC (Experimental): participants receiving efgartigimod PH20 SC on top of Prednisone
  Interventions: Biological: efgartigimod PH20 SC; Drug: Prednisone

INTERVENTIONS:
Biological: efgartigimod PH20 SC — Subcutaneous injection of efgartigimod coformulated with rHuPH20, a permeation enhancer
Drug: Prednisone — Oral Prednisone

SUMMARY:
The purpose of this study is to evaluate the safety of efgartigimod PH20 SC over a longer period of time in adult participants with moderate-to-severe bullous pemphigoid (BP) who have completed ARGX-113-2009 study. The study will also evaluate the efficacy of efgartigimod PH20 SC.

Eligible participants can roll over from the main study (ARGX-113-2009) to this open-label extension study (ARGX-113-2010). The study consists of a treatment period of up to 48 weeks in which participants receive efgartigimod PH20 SC. After the first 5 visits, the participants will visit the study centers at least once every 4 weeks. The participants who are not receiving efgartigimod PH20 SC (after the main study or currently on the study), will enter an observation period with study visits at least once every 8 weeks. If the participant relapses, they can re-enter the treatment period where they will receive efgartigimod PH20 SC. The treatment and observation period is followed by a follow-up period of 8 weeks. Oral or topical corticosterioids can be administered at the investigator's indiscretion

ELIGIBILITY:
Inclusion Criteria:

* Has completed the week 36 visit of ARGX-113-2009
* Is capable of providing signed informed consent and complying with protocol requirements
* Agrees to use contraceptive measures consistent with local regulations and the following: Women of childbearing potential must have a negative urine pregnancy test at baseline before receiving the study drug and must use one of the contraception methods described in the protocol from signing the ICF until the last dose of the study drug

Exclusion Criteria:

* Clinically significant disease, recent major surgery (within 3 months of baseline), or intends to have surgery during the study; or any other medical condition that, in the investigator's opinion would confound the results of the study or put the participant at undue risk
* Known hypersensitivity to the study drug or 1 of its excipients
* Permanently discontinued IMP in ARGX-113-2009 due to an adverse event (AE) considered related to the study drug and for whom the benefit/risk balance is not considered positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events, serious adverse events and adverse events of special interest | Up to 56 weeks
Rate of treatment discontinuation because of safety concerns | Up to 56 weeks
  Rate of treatment discontinuation because of safety concerns

SECONDARY OUTCOMES:
Proportion of participants achieving complete remission while off oral corticosteroids for ≥ 8 weeks | Up to 56 weeks
  Proportion of participants achieving complete remission while off oral corticosteroids for ≥ 8 weeks
Proportion of participants achieving complete remission or partial remission while off oral corticosteroids for ≥ 8 weeks | Up to 56 weeks
  Proportion of participants achieving complete remission or partial remission while off oral corticosteroids for ≥ 8 weeks
Proportion of participants achieving complete remission while on minimal oral corticosteroids therapy for ≥ 8 weeks | Up to 56 weeks
  Minimal oral corticosteroid therapy is defined as ≤0.10 mg/kg/day of prednisone (or an equivalent dose of another oral corticosteroid)
Proportion of participants achieving complete remission while off both oral corticosteroids and efgartigimod PH20 SC for ≥ 8 weeks | Up to 56 weeks
  Proportion of participants achieving complete remission while off both oral corticosteroids and efgartigimod PH20 SC for ≥ 8 weeks
Proportion of participants achieving complete remission or partial remission while off both oral corticosteroids and efgartigimod PH20 SC for ≥ 8 weeks | Up to 56 weeks
  Proportion of participants achieving complete remission or partial remission while off both oral corticosteroids and efgartigimod PH20 SC for ≥ 8 weeks
Duration of sustained remission | Up to 56 weeks
  Duration of sustained remission
Proportion of participants who relapse | Up to 56 weeks
  Proportion of participants who relapse
Time to relapse | Up to 56 weeks
  Time to relapse
Incidence of relapse | Up to 56 weeks
  Incidence of relapse
BPDAI activity scores over time | For participants not requiring treatment with efgartigimod PH20 SC at rollover: at weeks 0, 2, 4, 8, 16, 24, 32, 40, 48 and 56.
  The Bullous Pemphigoid Disease Area Index (BPDAI) is an internationally validated tool to objectively measure disease activity. The BPDAI differentiates scores for skin (erosions/blisters and urticaria/erythema) and mucous membrane activity in several anatomical locations
BPDAI activity scores over time | For participants continuing/starting efgartigimod PH20 SC treatment at rollover or relapse: at weeks 0, 2, 4 and 8 and then every 4 weeks until efgartigimod stop, every 8 weeks after efgartigimod stop and at weeks 48, 52 and 56.
  The Bullous Pemphigoid Disease Area Index (BPDAI) is an internationally validated tool to objectively measure disease activity. The BPDAI differentiates scores for skin (erosions/blisters and urticaria/erythema) and mucous membrane activity in several anatomical locations
IGA-BP scores over time | For participants not requiring treatment with efgartigimod PH20 SC at rollover: at weeks 0, 2, 4, 8, 16, 24, 32, 40, 48 and 56.
  The Investigator Global Assessment of Bullous Pemphigoid (IGA-BP) is a tool used to asses BP disease activity and severity. The IGA-BP categorizes the severity of BP on a numerical scale of 0 (clear) to 4 (severe).
IGA-BP scores over time | For participants continuing/starting efgartigimod PH20 SC treatment at rollover or relapse: at weeks 0, 2, 4 and 8 and then every 4 weeks until efgartigimod stop, every 8 weeks after efgartigimod stop and at weeks 48, 52 and 56.
  The Investigator Global Assessment of Bullous Pemphigoid (IGA-BP) is a tool used to asses BP disease activity and severity. The IGA-BP categorizes the severity of BP on a numerical scale of 0 (clear) to 4 (severe).
Itch NRS over time | For participants not requiring treatment with efgartigimod PH20 SC at rollover: at weeks 0, 2, 4, 8, 16, 24, 32, 40, 48 and 56.
  The Itch Numerical Rating Scale (NRS) is used to indicate pruritic symptoms of BP. The score varies between 0 (best outcome) to 10 (worst outcome)
Itch NRS over time | For participants continuing/starting efgartigimod PH20 SC treatment at rollover or relapse: at weeks 0, 2, 4 and 8 and then every 4 weeks until efgartigimod stop, every 8 weeks after efgartigimod stop and at weeks 48, 52 and 56.
  The Itch Numerical Rating Scale (NRS) is used to indicate pruritic symptoms of BP. The score varies between 0 (best outcome) to 10 (worst outcome)
Rate of treatment failure | Up to 56 weeks
  Rate of treatment failure
Glucocorticoid Toxicity Index (GTI)-related scores, including the Glucocorticoid Toxicity Index - Aggregate Improvement Score (GTI-AIS) over time | For participants not requiring treatment with efgartigimod PH20 SC at rollover: at weeks 0, 24 and 48.
  Glucocorticoid Toxicity Index (GTI)-related scores, including the Glucocorticoid Toxicity Index - Aggregate Improvement Score (GTI-AIS) over time
Glucocorticoid Toxicity Index (GTI)-related scores, including the Glucocorticoid Toxicity Index - Aggregate Improvement Score (GTI-AIS) over time | For participants continuing/starting efgartigimod treatment at rollover or relapse: weeks 0, 8, every 16 weeks until and after efgartigimod treatment stop and at week 48.
  Glucocorticoid Toxicity Index (GTI)-related scores, including the Glucocorticoid Toxicity Index - Aggregate Improvement Score (GTI-AIS) over time
Glucocorticoid Toxicity Index (GTI)-related scores, including the Glucocorticoid Toxicity Index Cumulative Worsening Score (GTI-CWS) over time | For participants not requiring treatment with efgartigimod PH20 SC at rollover: at weeks 0, 24 and 48.
  Glucocorticoid Toxicity Index (GTI)-related scores, including the Glucocorticoid Toxicity Index Cumulative Worsening Score (GTI-CWS) over time
Glucocorticoid Toxicity Index (GTI)-related scores, including the Glucocorticoid Toxicity Index Cumulative Worsening Score (GTI-CWS) over time | For participants continuing/starting efgartigimod treatment at rollover or relapse: weeks 0, 8, every 16 weeks until and after efgartigimod treatment stop and at week 48.
  Glucocorticoid Toxicity Index (GTI)-related scores, including the Glucocorticoid Toxicity Index Cumulative Worsening Score (GTI-CWS) over time
Glucocorticoid Toxicity Index (GTI)-related scores, including the Glucocorticoid Toxicity Index Specific List (GTI-SL) over time | For participants not requiring treatment with efgartigimod at rollover: at weeks 0, 24 and 48.
  Glucocorticoid Toxicity Index (GTI)-related scores, including the Glucocorticoid Toxicity Index Specific List (GTI-SL) over time
Glucocorticoid Toxicity Index (GTI)-related scores, including the Glucocorticoid Toxicity Index Specific List (GTI-SL) over time | For participants continuing/starting efgartigimod treatment at rollover or relapse: weeks 0, 8, every 16 weeks until and after efgartigimod treatment stop and at week 48.
  Glucocorticoid Toxicity Index (GTI)-related scores, including the Glucocorticoid Toxicity Index Specific List (GTI-SL) over time
EQ-5D-5L scores over time | For participants not requiring treatment with efgartigimod PH20 SC at rollover: at weeks 0, 24 and 48.
  The EQ-5D-5L questionnaire is a patient-reported outcome measure, ranging 0 to 100 (lower score, worse outcome).
EQ-5D-5L scores over time | For participants continuing/starting efgartigimod treatment at rollover or relapse: at weeks 0, 8, every 16 weeks until and after efgartigimod PH20 SC treatment stop and at week 48.
  The EQ-5D-5L questionnaire is a patient-reported outcome measure, ranging 0 to 100 (lower score, worse outcome).
ABQoL scores over time | For participants not requiring treatment with efgartigimod PH20 SC at rollover: at weeks 0, 24 and 48.
  The Autoimmune Bullous Disease Quality of Life (ABQoL) was developed and validated for determining the impact of AIBDs and their therapies on the daily lives of patients.
ABQoL scores over time | For participants continuing/starting efgartigimod treatment at rollover or relapse: at weeks 0, 8, every 16 weeks until and after efgartigimod PH20 SC treatment stop and at week 48.
  The Autoimmune Bullous Disease Quality of Life (ABQoL) was developed and validated for determining the impact of AIBDs and their therapies on the daily lives of patients.
DLQI scores over time | For participants not requiring treatment with efgartigimod PH20 SC at rollover: at weeks 0, 24 and 48.
  The Dermatology Life Quality Index (DLQI) consists of 10 questions concerning the participant's perception of the impact of skin diseases on different aspects of their health-related QoL the previous week. The impact of each aspect on the QoL assessment is scored qualitatively, ranging from "not at all" to "very much."
DLQI scores over time | For participants continuing/starting efgartigimod treatment at rollover or relapse: at weeks 0, 8, every 16 weeks until and after efgartigimod PH20 SC treatment stop and at week 48.
  The Dermatology Life Quality Index (DLQI) consists of 10 questions concerning the participant's perception of the impact of skin diseases on different aspects of their health-related QoL the previous week. The impact of each aspect on the QoL assessment is scored qualitatively, ranging from "not at all" to "very much."
Percent changes from baseline over time for anti-BP180 and anti-BP-230 antibody levels | For participants not requiring treatment with efgartigimod PH20 SC at rollover: at weeks 0, 2, 4, 8, 16, 24, 32, 40, 48 and 56.
  Percent changes from baseline over time for anti-BP180 and anti-BP-230 antibody levels
Percent changes from baseline over time for anti-BP180 and anti-BP-230 antibody levels | For participants continuing/starting efgartigimod PH20 SC treatment at rollover or relapse: at weeks 0, 2, 4 and 8 and then every 4 weeks to efgartigimod stop, every 8 weeks after efgartigimod stop and at weeks 48, 52 and 56.
  Percent changes from baseline over time for anti-BP180 and anti-BP-230 antibody levels
Incidence of antidrug antibody(ies) (ADA) against efgartigimod (serum levels) | For participants not requiring treatment with efgartigimod PH20 SC at rollover: at weeks 0, 4, 8, 16, 24, 32, 40, 48 and 56.
  Incidence of antidrug antibody(ies) (ADA) against efgartigimod (serum levels)
Incidence of antidrug antibody(ies) (ADA) against efgartigimod (serum levels) | For participants continuing/starting efgartigimod treatment at rollover or relapse: at weeks 0, 2, 4 and 8 and then every 8 weeks until and after efgartigimod PH20 SC stop and at weeks 48, 52 and 56.
  Incidence of antidrug antibody(ies) (ADA) against efgartigimod (serum levels)

CONTACTS AND LOCATIONS:
Locations (40):
- United States (6):
  - Medical Dermatology Specialists, Phoenix, Arizona
  - First OC Dermatology, Fountain Valley, California
  - Miami Dermatology and Laser Institute, Miami, Florida
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Saint Louis University, St Louis, Missouri
  - Wright State Physicians, Fairborn, Ohio
- Premier Specialists, Kogarah, Australia
- Diagnostic and Consulting Center Aleksandrovska EOOD, Sofia, Bulgaria
- China (3):
  - West China Hospital of Sichuan University, Chengdu
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai
- Poliklinika Solmed, Zagreb, Croatia
- Fakultni nemocnice Bulovka, Prague, Czechia
- Germany (6):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Carl Gustav Carus an der TU Dresden, Dresden
  - Universitatsklinikum Dusseldorf, Düsseldorf
  - Universitatsklinikum Schleswig-Holstein, Kiel
  - LMU Klinikum der Universität, München
  - Universitätsklinikum Würzburg, Würzburg
- Greece (2):
  - Hospital of Venereal and Skin Diseases A.Syggros, Athens
  - Hospital Of Skin And Venereal Diseases of Thessaloniki, Thessaloniki
- Semmelweis Egyetem, Budapest, Hungary
- Sheba Medical Center - PPDS, Ramat Gan, Israel
- Italy (8):
  - Azienda Ospedaliero Universitaria Policlinico Vittorio Emanuele, Catania
  - Azienda USL Toscana Centro - Ospidale Piero Palagi, Florence
  - Azienda Sanitaria Di Firenze, Florence
  - Ospedale Policlinico San Martino, Genova
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
  - Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia
  - IDI IRCCS - Istituto Dermopatico dell'Immacolata, Roma
  - Fondazione Policlinico Universitario A. Gemelli, Rome
- Hokkaido University Hospital, Sapporo, Japan
- Universitair Medisch Centrum Groningen, Groningen, Netherlands
- University Clinical Center of Serbia - PPDS, Belgrade, Serbia
- Slovakia (2):
  - Univerzitna nemocnica Bratislava, Bratislava
  - Fakultna nemocnica Trnava, Trnava
- Spain (3):
  - Hospital Universitario Clínico San Cecilio, Granada
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Doctor Peset, Valencia
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom